CLINICAL TRIAL: NCT06186999
Title: Social and Demographic Determinants of Fatigue in Patients With Inflammatory Bowel Disease in Remission
Acronym: SOFA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01692-43
Record Dates: First submitted 2023-10-13; First posted 2024-01-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Remission; Fatigue
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to identify the social and demographic determinants of fatigue in patients with inflammatory bowel disease in remission.

Secondly, the objectives of the study are to:

* Assess the impact of fatigue on the quality of life of patients with inflammatory bowel disease in remission.
* To determine the profile of patients with inflammatory bowel disease in remission who are fatigued.

To this end, during a consultation or hospitalization, participants will be asked to respond independently to various questionnaires (FACIT-F, DIPCare, SSQ6, questionnaire on socio-demographic determinants and IBD disk). Characteristics of the type of chronic inflammatory bowel disease will be collected from medical records.

There will be no patient follow-up as part of the study. Participants may be contacted by telephone by the center's investigator within 2 weeks of the interview in the event of a partial or imprecise response.

ELIGIBILITY:
Inclusion Criteria:

* Patient in clinical remission for at least 6 months:

  * for Crohn's disease patients: Harvey Bradshaw Index (HBI) score ≤ 4
  * for patients with ulcerative colitis: a partial Mayo score (PMS) ≤ 2 with each subscore of 1 or less)
* Patient in biological remission for at least 6 months fecal calprotectin <250 μg/g and CRP <5 mg/
* Documented diagnosis of Crohn's disease or ulcerative colitis based on standard clinical, endoscopic and histological criteria
* FACIT-F score < 40 (defining significant fatigue)
* Subjects at least 18 years of age at the time of study inclusion

Exclusion Criteria:

* Severe acute colitis
* Active infection with HIV, hepatitis B, hepatitis C, or untreated tuberculosis
* Patient(s) objecting to the use of their data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns patients with chronic inflammatory bowel disease in remission, such as Crohn's disease or ulcerative colitis.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Description of the relationship : fatigue - social precariousness | at enrollment
  Description of the relationship between social precariousness assessed by the "DiPCare" questionnaire and fatigue assessed by the FACIT-F questionnaire in patients with inflammatory bowel disease in remission.
Description of the relationship : patient social support - fatigue. | at enrollment
  Description of the relationship between patient social support (availability and satisfaction of the patient's entourage) assessed by the "SARASON" (or "SSQ6") questionnaire and fatigue assessed by the FACIT-F questionnaire in patients with inflammatory bowel disease in remission.
Description of the relationship : demographic determinants - fatigue. | at enrollment
  Description of the relationship between demographic determinants assessed by the questionnaire, and fatigue assessed by the FACIT-F questionnaire in patients with inflammatory bowel disease in remission.

SECONDARY OUTCOMES:
Assessing quality of life in IBD patients | at enrollment
  Functional visual handicap score based on IBD-Disk visual aid, evaluated at enrollment.

OTHER OUTCOMES:
Caracterization of patients with chronic bowel disease (IBD) in remission in function of anthropometric and clinical parameters. | at enrollment
  Descriptif analysis of IBD patients according to socio demographic and health caracteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Mathieu, Pr, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - CHU Bordeaux Hôpital Haut Lévêque, Bordeaux
  - CHUGA, Grenoble
  - Chu Lyon Sud _ Hcl, Lyon
  - Chu Montpellier, Montpellier